CLINICAL TRIAL: NCT00279461
Title: Vitamin D Deficiency Causes Immune Dysfunction and Enables or Perpetuates the Development of Rheumatoid Arthritis: Clinical Trial and Investigations on Dendritic Cells
Brief Title: Vitamin D Deficiency Causes Immune Dysfunction and Enables or Perpetuates the Development of Rheumatoid Arthritis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Dr. Levy terminated from IU in December 2009. Indiana University has no record that this study was initiated prior to his termination.
Sponsor: Indiana University (Other)
Responsible Party: Ernesto N Levy, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21562; No secondary ID at this time
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Arthritis, Rheumatoid; Vitamin D Deficiency
Keywords: Rheumatoid Arthritis; Vitamin D
MeSH Terms: conditions — Arthritis, Rheumatoid; Vitamin D Deficiency | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A, (Experimental): Arm A: Vitamin D 2,000 units daily all in one capsule for 6 months
  Interventions: Drug: Placebo in arm A and Vitamin D in arm B
- B (Placebo Comparator): Arm B: matching placebo one capsule daily for 6 months
  Interventions: Drug: vitamin D 3 for arm A ,and matching placebo for arm B

INTERVENTIONS:
Drug: Placebo in arm A and Vitamin D in arm B — Vitamin D3 at 2,000 units daily, all in one capsule, for 6 months and Placebo provided in matching capsule, one capsule daily, for 6 months
  Other Names: Vitamin D3 is also called cholecalciferol
  Arms: A,
Drug: vitamin D 3 for arm A ,and matching placebo for arm B — Arm A 2,000 units of Vitamin D3 in one capsule daily for 6 months. Arm B matching placebo capsule, one daily for 6 months
  Other Names: Cholecalciferol
  Arms: B

SUMMARY:
Recent studies have demonstrated that subjects with low blood levels of vitamin D are at a higher risk of developing autoimmune diseases such as Rheumatoid Arthritis (RA). We are pursuing these studies to test the hypothesis that restoration of vitamin D levels ameliorates the manifestations of RA. We will test this hypothesis by inviting patients with RA to participate in a trial that examines the effects of oral vitamin D administration on the clinical expression of this disease. For this purpose, the participants of this trial will be asked to take an oral dose of 2,000 units of vitamin D daily for 6 months. We will examine the participant's joints, assess disease activity measures, and determine his/her blood levels of vitamin D before starting this treatment and periodically thereafter.

DETAILED DESCRIPTION:
Rationale : Low vitamin D levels hinders the ability of the macrophage to produce activated 1-25Dihydroxyvitamin at sites of inflammation. 1-25Dihydroxyvitamin D has important immunoregulatory functions including down-regulation of antigen-presenting cells such as dendritic cells. Under the influence of 1-25Dihydroxyvitamin D, these dendritic cells become tolerogenic - as opposed to immunogenic - and abrogate an immune response at early stages. Immunogenic dendritic cells play a key role in the development of autoimmune diseases such as Rheumatoid Arthritis (RA) by "presenting" self-antigens to the immune system. Vitamin D levels are frequently low in patients with RA. Restoring vitamin D availability to normal levels in patients with RA may induce improvement of disease manifestations through expansion of the tolerogenic dendritic cell subset.

Key Objectives:

* Conduct a double-blind randomized clinical trial, to test the hypothesis that vitamin D administered to patients with active RA has beneficial effects on this disease.
* Determine if vitamin D administered to patients with RA. induces expansion of the tolerogenic dendritic cell subset by analyzing patterns of cell surface marker expression on dendritic cells at different time points during the clinical trial (translational studies).

Study Population: We will recruit early RA patients (not more that 12 month duration of disease)with active joint inflammation cared for at this institution.Participants must be subjects with active RA at the time of inclusion, who are 18 years of age or older and have no history of other autoimmune disorders or other disorders such as cancer or osteoporosis which are also linked to vitamin D deficiency. The eligible patients with active RA should be on treatment for RA with Methotrexate at the time of inclusion. Patients taking anti-cytokine treatments (considered not standard) would be excluded. Other exclusions include hypercalcemia, and a history of renal failure or renal stones.

20-25 participants will be allocated to the Vitamin D Group, Arm A. 20-25 participants will be allocated to Placebo Group Arm B Allocation will be conducted in a randomized, double-blind fashion.

Summary of Procedures : After signing a written consent, all potential candidates will undergo a screening interview with the PI and screening blood tests (a blood sample of 20 ml is required).

RA subjects who qualify to receive the study treatment will be randomized to receive oral vitamin D 2,000 units or placebo daily for 6 months. Patients will be examined on a monthly basis and will be drawn a 20 ml blood sample every 2 months for monitoring purposes for a period of 12 month. The participants within the clinical trial who also participate in the translational studies on dendritic cells, will be drawn an additional blood sample of 40 ml on the first month and at the end of the study to isolate their blood dendritic cells. We will study the expression of different activation markers on dendritic cells from consenting participants using various immunologic techniques. This will allow us to identify and quantify the tolerogenic dendritic cells..

ELIGIBILITY:
Inclusion Criteria:

This study will involve two groups of patients fulfilling the following eligibility requirements:

* they should have early (not more than 12 month duration) active RA as determined by the diagnostic criteria and active status definitions as described below, and
* they should have at the time of inclusion a 25(OH)vitamin D level below 30 ng/ml.
* All RA patients in this study will satisfy the American Rheumatism Association 1987 revised criteria for the diagnosis of RA. Active disease will be defined by the presence of at least 3 swollen joints, ≥6 tender or painful joints and at least 2 of the following features: duration of morning stiffness 60 minutes, erythrocyte sedimentation rate (ESR) ≥28 mm/hour and serum CRP level of at least 2.0 mg/dl (26).
* Only research subjects of either gender who are 18 years of age or older will be invited to participate.
* One group, Group A, will include active RA patients receiving treatment with methotrexate. A concomitant prescription of non-steroidal anti-inflammatory drugs (NSAIDs), and/or Prednisone ≤ 10 mg/day will be allowed. Treatment with anti-TNF agents, Abatacept or other immunosuppressives constitute exclusion criteria.
* To minimize the impact of pre-existing treatments on the final outcome of this trial, patients taking NSAIDs and/or prednisone will be required to receive unchanged doses of these medications for at least 1 month. No modifications of these treatments will be allowed during the study. In addition to their methotrexate treatment, patients within Group A will receive placebo every day for 12 consecutive months.
* The second group, Group B, will include those patients as described for Group A who instead of placebo will receive oral vitamin D, 1,000 units every day for 12 consecutive months added to their standard RA treatment.

Exclusion Criteria:

* Because cancer and other autoimmune diseases may be more frequent in individuals with a moderate deficiency of vitamin D, subjects with a history of these conditions will be excluded. Because of the remote possibility of vitamin D-induced hypercalcemia, we are aiming at recruiting patients with RA who are otherwise healthy. We will exclude patients who in the past had or currently have cancer (except if considered cured), kidney stones, chronic renal failure, congestive heart failure, arrythmia requiring treatment with antiarrythmics, pulmonary conditions requiring ambulatory oxygen, abnormal levels of calcium or elevated PTH.
* Patients who use Digoxin (drug interaction), or had experienced angina or myocardial infarction in the last 3 years also will be excluded, but patients whose coronary artery disease has been asymptomatic for at least 3 years and who do not have congestive heart failure will be allowed to participate.
* Patients who develop hypercalcemia, kidney stones, elevation of 25(OH)vitamin D> 90 ng/ml also will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
ACR20 | Baseline and every 2 months for 6 months

SECONDARY OUTCOMES:
Changes in surface marker expression of blood myeloid dendritic cells | Baseline and at completion of study on the 6th month

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto N Levy, MD, Principal Investigator — India na University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Andjelkovic Z, Vojinovic J, Pejnovic N, Popovic M, Dujic A, Mitrovic D, Pavlica L, Stefanovic D. Disease modifying and immunomodulatory effects of high dose 1 alpha (OH) D3 in rheumatoid arthritis patients. Clin Exp Rheumatol. 1999 Jul-Aug;17(4):453-6. PMID 10464556
- [Background] Cantorna MT, Hayes CE, DeLuca HF. 1,25-Dihydroxycholecalciferol inhibits the progression of arthritis in murine models of human arthritis. J Nutr. 1998 Jan;128(1):68-72. doi: 10.1093/jn/128.1.68. PMID 9430604
- [Background] Adorini L, Penna G, Giarratana N, Roncari A, Amuchastegui S, Daniel KC, Uskokovic M. Dendritic cells as key targets for immunomodulation by Vitamin D receptor ligands. J Steroid Biochem Mol Biol. 2004 May;89-90(1-5):437-41. doi: 10.1016/j.jsbmb.2004.03.013. PMID 15225816